CLINICAL TRIAL: NCT02322619
Title: An Open Label, Balanced, Randomized, Two-treatment, Two-period, Two-sequence, Single Dose, Crossover, Oral Bioequivalence Study of Moxifloxacin Tablets, 400 mg of Dr. Reddy's Laboratories Limited, Comparing With Avelox® Tablets 400 mg of Bayer Healthcare Pharmaceuticals Inc. in Healthy, Adult Human Subjects Under Fasting Conditions
Brief Title: Bio-equivalency Study of Moxifloxacin Tablets, 400 mg Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 054-12
Record Dates: First submitted 2014-12-18; First posted 2014-12-23 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Healthy
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Moxifloxacin Tablets 400 mg (Experimental): Moxifloxacin Tablets 400 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Moxifloxacin Tablets 400 mg
- Avelox Tablets 400 mg (Active Comparator): Avelox® Tablets 400 mg of Bayer Healthcare Pharmaceuticals Inc.
  Interventions: Drug: Moxifloxacin Tablets 400 mg

INTERVENTIONS:
Drug: Moxifloxacin Tablets 400 mg — Moxifloxacin Tablets 400 mg of Dr. Reddy's Laboratories Limited
  Other Names: Avelox

SUMMARY:
An open label, balanced, randomized, two-treatment, two-period, two-sequence, single dose, crossover, oral bioequivalence study in human subjects under fasting conditions.

DETAILED DESCRIPTION:
An open label, balanced, randomized, two-treatment, two-period, two-sequence, single dose, crossover, oral bioequivalence study of moxifloxacin tablets 400 mg of Dr. Reddy's Laboratories Limited, comparing with Avelox ® Tablets 400 mg of Bayer Healthcare Pharmaceuticals Inc. in healthy, adult, human subjects under fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult human volunteers between 18 to 45 years of age (both inclusive) living in and around Ahmedabad city or western part of India.
* Having a Body Mass Index (BMI) between 18.5 to 24.9 (both inclusive), calculated as weight in kg / height in m2.

Not having any significant diseases or clinically significant abnormal findings during screening, medical history, clinical examination, laboratory evaluations, 12- lead ECG and X-ray chest (postero-anterior view) recordings.

* Able to understand and comply with the study procedures, in the opinion of the investigator.
* Able to give voluntary written informed consent for participation in the trial.
* In case of female subjects:

  * Surgically sterilized at least 6 months prior to study participation or
  * If of child bearing potential is willing to use a suitable and effective double barrier contraceptive method or intra uterine device during the study. and
  * Pregnancy test must be negative.

Exclusion Criteria:

* Known hypersensitivity or idiosyncratic reaction to Moxifloxacin, other Quinolones or any of the excipients or any related drug.
* History or presence of any disease or disorder known to influence bone metabolism, compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
* Ingestion of medicine [including vitamin, herbal supplements and any enzyme modifying drugs, including strong inhibitors of cytochrome P450 (CYP) enzymes and strong inducers of CYP enzymes] at any time within 14 days prior to check in of period-I. In any such case subject selection will be at the discretion of the Principal Investigator.
* If the QTc interval will be more than 450 ms on ECG measurement at the time of screening.
* Any history or presence of hypokalamia, QT prolongation including torsades de pointe.
* Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or NSAIDs induced urticaria.
* A recent history of harmful use of alcohol(less than 2 years), i.e. alcohol consumption of more than 14 standard drinks per week for men and more than 7 standard drinks per week for women (A standard drink is defined as 360 ml of beer or 150 ml of wine or 45 ml of 40% distilled spirits, such as rum, whisky, brandy etc) or consumption of alcohol or alcoholic products within 48 hours prior to check in.
* Smokers, who smoke 10 or more than 10 cigarettes / day or inability to abstain from smoking during the study.
* The presence of clinically significant abnormal laboratory values during screening.
* Use of any recreational drugs or history of drug addiction or testing positive in pre study drug scans.
* History or presence of psychiatric disorders.
* A history of difficulty with donating blood.
* Donation of blood (1 unit or 350 mL) or receipt of an investigational medicinal product or participation in a drug research study within 90 days prior to receiving the first dose of study medicine.

Note: In case the blood loss was less than or equal to 200 mL; subject may be enrolled 60 days after blood donation or after the last sample of previous study

* A positive hepatitis screen including hepatitis B surface antigen and/or HCV antibodies.
* A positive test result for HIV antibody.
* Consumption of grape fruit or grape fruit products within 48 hours prior to check in.
* An unusual diet, for whatever reason (e.g. low-sodium), for four weeks prior to check in of Period I. In any such case subject selection will be at the discretion of the Principal Investigator.
* Nursing mothers (females).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Area under curve | 0.167, 0.333, 0.500, 0.750, 1.000, 1.333, 1.667, 2.000, 2.333, 2.667, 3.000, 3.500, 4.000, 4.500, 5.000, 6.000, 8.000, 10.000, 12.000, 16.000, 24.000, 36.000 and 48.000 post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Shashikanth Sharma, MD, Principal Investigator — Lambda Therapeutic Research Ltd.